CLINICAL TRIAL: NCT02243839
Title: Thrombolytic Therapy Versus Surgery for Obstructive Prosthetic Valve Thrombosis: A Randomized Multicenter Study
Brief Title: Thrombolytic Therapy Versus Surgery for Obstructive Prosthetic Valve Thrombosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, MEHMET OZKAN, Professor, Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KOSUYOLU3
Record Dates: First submitted 2014-09-12; First posted 2014-09-18 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Obstructive Thrombus
Keywords: Prosthetic valve; Thrombosis; Surgery; Thrombolytic therapy; Transesophageal echocardiography
MeSH Terms: conditions — Thrombosis | interventions — Thrombolytic Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thrombolytic therapy (Active Comparator): In the first arm, thrombolytic therapy (TT) is performed to the patients with obstructive prosthetic valve thrombosis. The TT regimen depends on the functional status of the patient. In patients with NYHA class III-IV dyspnea low dose, relatively faster TT regimen (25 mg tPA/6 hours) is performed. In patients with NYHA class I-II dyspnea TT with low dose and ultra-slow infusion of tPA (25 mg tPA/25 hours) is performed. During TT, patients are followed up with transesophageal echocardiography in every 24 hours.
  Interventions: Drug: Thrombolytic Therapy
- Surgery (Active Comparator): In the second arm, redo valve surgery is performed for obstructive valve thrombosis. Intraoperative and postoperative results are recorded
  Interventions: Procedure: Surgery

INTERVENTIONS:
Drug: Thrombolytic Therapy — Thrombolytic therapy is performed to the patients with obstructive prosthetic valve thrombosis
  Arms: Thrombolytic therapy
Procedure: Surgery — Redo valve surgery is performed for obstructive valve thrombosis
  Arms: Surgery

SUMMARY:
Prosthetic heart valve thrombosis is a serious complication with high mortality and morbidity The best treatment of PVT is controversial, although surgery and thrombolysis options have been available. In this randomized and multicenter study, the investigators compared thrombolytic therapy versus surgery for the treatment of patients with obstructive prosthetic valve thrombosis.

DETAILED DESCRIPTION:
Two different randomization group have been defined and patients with obstructive prosthetic valve thrombosis are included in each group randomly. In the first arm, thrombolytic therapy (TT) is performed to the patients with obstructive prosthetic valve thrombosis. The TT regimen depends on the functional status of the patient. In patients with NYHA class III-IV dyspnea low dose, relatively faster TT regimen (25 mg tPA/6 hours) is performed. In patients with NYHA class I-II dyspnea TT with low dose and ultra slow infusion of tPA (25 mg tPA/25 hours) is performed. During TT, patients are followed up with transesophageal echocardiography in every 24 hours. In the second arm, redo valve surgery is performed for obstructive valve thrombosis. This multicenter study is conducted in Cardiology and Cardiovascular Surgery Departments of Kosuyolu Kartal Heart Training and Research Hospital, Istanbul, Turkey, Siyami Ersek Heart Training and Research Hospital, Istanbul, Turkey, Ankara Heart Training and Research Hospital, Ankara, Turkey, İzmir Atatürk Heart Training and Research Hospital, İzmir, Turkey, Erzurum Atatürk University Faculty of Medicine, Erzurum, Turkey, Diyarbakır Dicle University Faculty of Medicine, Diyarbakır, Turkey and Kars Kafkas University Faculty of Medicine, Kars, Turkey. Informed consent is taken from all patients.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive prosthetic valve thrombosis

Exclusion Criteria:

* Non-obstructive prosthetic valve thrombosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Thrombolytic success | Up to 10 days
  In the absence of fatal or nonfatal major complications;
  Obstructive thrombus:
  Doppler documentation of the resolution of increased gradient and decreased valve area.
  Clinical improvement in symptoms. Reduction by ≥75% in major diameter or area of the thrombus. Complete success was defined when all 3 criteria were met and partial success was defined as less than 3
  Nonobstrucive thrombus:
  Complete success: ≥75% reduction in thrombus area. Partial success: 50%-75% reduction in thrombus area
Non-fatal complications for thrombolytic therapy | Participants will be followed for the duration of hospital stay, an expected average of 3 weeks
  Nonfatal major complication: Ischemic stroke, intracranial hemorrhage, embolism (coronary or peripheral), bleeding requiring transfusion.
  Nonfatal minor complication: Bleeding without need for transfusion, TIA.
Successful Surgery | Participants will be followed for the duration of hospital stay, an expected average of 3 weeks; and postoperative 3 months
  Successful redo valve surgery in the absence of fatal and non fatal major complications.
Complications for surgery | Participants will be followed for the duration of hospital stay an expected average of 3 weeks; and postoperative 3 month
  Non fatal major complications: Ischemic stroke, intracranial hemorrhage, embolism (coronary or peripheral), bleeding requiring transfusion, pericardial tamponade, sepsis, pacemaker requirement, mediastinitis, wound infections, acute renal failure Minor complications: bleeding requiring transfusion, plevral effusion, pericardial effusion without tamponade
In hospital mortality | Participants will be followed for the duration of hospital stay, an expected average of 3 weeks
  All cause in-hospital mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Kosuyolu Kartal Heart Training and Research Hospital, Istanbul, Turkey (Türkiye)